CLINICAL TRIAL: NCT02429843
Title: A Phase 1B Dose-Escalation Study of TRC105 in Combination With Paclitaxel/Carboplatin and Bevacizumab in Patients With Stage 4 Non-Squamous Cell Lung Cancer
Brief Title: A Study of TRC105 in Combination With Paclitaxel/Carboplatin and Bevacizumab in Non-Squamous Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Principal Investigator, Francisco Robert,MD, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F150128005 (UAB 1504)
Record Dates: First submitted 2015-03-18; First posted 2015-04-29 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Lung Cancer
Keywords: Non-squamous cell lung cancer; Non-squamous non-small cell lung cancer; vascular endothelial growth factor (VEGF); TRC105
MeSH Terms: conditions — Lung Neoplasms | interventions — carotuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Standard treatment + TRC105 (Experimental): In addition to standard treatment of paclitaxel, carboplatin, and bevacizumab, dosing of TRC105 will begin at 8 mg/kg. However a lower dose level has also been included (6 mg/kg) and will be enrolled if 8 mg/kg is found to exceed the maximum tolerated dose. Following the appropriate pre-medication regimen, the first weekly TRC105 dose (cycle 1 day 8) will be split into two doses whereby 3 mg/kg is administered on cycle 1 day 8 and the balance (e.g., 5 mg/kg for Dose Level 1) is administered on cycle 1 day 11. Beginning with cycle 1 day 15 and thereafter, the full TRC105 dose will be administered intravenously each week during the 21-day cycle. Intra-patient dose reductions are allowed beginning in cycle 2.
  Interventions: Drug: TRC105

INTERVENTIONS:
Drug: TRC105 — Each patient will be dosed with 6, 8, or 10 mg/kg of TRC105 up to a maximum dose of 850 mg for women and 1,000 mg for men based upon overall body weight.

SUMMARY:
This is a single center, open-label, nonrandomized, phase 1b study of TRC105 in combination with standard dose treatment in patients with stage IV non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
Advanced non-small cell lung cancer has been historically difficult to treat, and novel agents are in dire need.TRC105 has been shown to enhance the anti-angiogenic effect of bevacizumab and may result in more effective angiogenesis inhibition and improved clinical efficacy when combined with bevacizumab and paclitaxel/carboplatin. Participants will be treated with the combination drugs for 6 cycles of therapy (3 weeks per cycle) and may or may not be placed on maintenance therapy depending upon the induction response. Maintenance therapy will continue until there is disease progression, unacceptable toxicity, or patient withdrawal. Blood collections and tumor assessments will be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve, stage 4 Non-Squamous Cell Lung Cancer
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST).
* Age of 19 years or older.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
* Resolution of all acute adverse events resulting from prior cancer therapies to NCI Common Terminology Criteria for Adverse Events (CTCAE) grade ≤1 or baseline (except alopecia or neuropathy).
* Adequate organ function as defined by the following criteria:
* Serum aspartate transaminase (AST; serum glutamate oxaloacetate transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamate pyruvate transaminase [SGPT]) ≤2.5 x upper limit of normal (ULN) or ≤5 x ULN in cases of liver metastases.
* Total serum bilirubin ≤1.5 times the upper limit of normal.
* Absolute neutrophil count (ANC) ≥1500/μL.
* Platelets ≥100,000/μL without transfusion support within the past 28 days.
* Hemoglobin ≥9.0 g/dL without transfusion support within the past 28 days (erythropoietin or darbepoietin permitted).
* Serum creatinine ≤1.5 times the upper limit of normal or creatinine clearance >30 mL/min by Cockcroft-Gault formula.
* International Normalized Ratio (INR) from 0.8 to 1.2.
* Willingness and ability to consent for self to participate in study.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Non-small cell lung cancer of squamous histology.
* Prior treatment with TRC105.
* Current treatment on another therapeutic clinical trial.
* Receipt of a small molecule anticancer agent, including an investigational anticancer small molecule, within 14 days of starting study treatment.
* Receipt of a large molecule anticancer agent (e.g., antibody), including an investigational anticancer antibody, within 28 days of starting study treatment.
* No major surgical procedure or significant traumatic injury within 6 weeks prior to study registration, and must have fully recovered from any such procedure; date of surgery (if applicable) or the anticipated need for a major surgical procedure within the next six months. The following are not considered to be major procedures and are permitted up to 7 days before therapy initiation: thoracentesis, paracentesis, port placement, laparoscopy, thorascopy, tube thoracostomy, bronchoscopy, endoscopic ultrasonographic procedures, mediastinoscopy, skin biopsies, incisional biopsies, imaging-guided biopsy for diagnostic purposes, and routine dental procedures.
* Patients who have received wide field radiotherapy ≤28 days (defined as >50% of volume of pelvic bones or equivalent) or limited field radiation for palliation <14 days prior to study registration or those patients who have not recovered adequately from side effects of such therapy.
* Uncontrolled chronic hypertension defined as systolic >150 or diastolic >90 despite optimal therapy (initiation or adjustment of BP medication prior to study entry is allowed provided that the average of 3 BP readings at a visit prior to enrollment is <140/90 mm Hg).
* History of brain involvement with cancer, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease. Patients with radiated or resected lesions are permitted, provided the lesions are fully treated and inactive, patients are asymptomatic, and no steroids have been administered for at least 28 days.
* Angina, myocardial ischemia (MI), symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG) within the past 6 months. Deep venous thrombosis within 6 months, unless the patient is anticoagulated without the use of warfarin for at least 2 weeks. In this situation, low molecular weight heparin is preferred.
* Active bleeding or pathologic condition that carries a high risk of bleeding (e.g. hereditary hemorrhagic telangiectasia). Patients who have been uneventfully anticoagulated with low molecular weight heparin are eligible.
* Thrombolytic use (except to maintain i.v. catheters) or anticoagulant use within 10 days prior to first day of study therapy.
* Cardiac dysrhythmias of NCI CTCAE grade ≥2 within the last 28 days.
* Known active viral or nonviral hepatitis or cirrhosis.
* History of hemorrhage or hemoptysis (>½ teaspoon bright red blood) within 3 months of starting study treatment.
* History of peptic ulcer disease or erosive gastritis within the past 3 months, unless treated for the condition and complete resolution has been documented by esophagogastroduodenoscopy (EGD) within 28 days of starting study treatment.
* History of gastrointestinal perforation or fistula in the past 6 months, or while previously on antiangiogenic therapy, unless underlying risk has been resolved (e.g., through surgical resection or repair).
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness.
* Pregnancy or breastfeeding. Female patients must be surgically sterile (i.e.: hysterectomy) or be postmenopausal, or must agree to use effective contraception during the study and for 3 months following last dose of TRC105. All female patients of reproductive potential must have a negative pregnancy test (serum or urine) within 7 days prior to first dose. Male patients must be surgically sterile or must agree to use effective contraception during the study and for 3 months following last dose of TRC105.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with a change in medical management | Baseline up to 28 days after the last cycle
  Adverse events will be graded using the NCI Common Terminology for Criteria for Adverse Events(CTCAE). Incidence, timing, and relatedness of adverse events will be considered as factors in the change of a patient's medical management.

SECONDARY OUTCOMES:
Measurement of tumor response | Baseline to 3 years
  Radiological tumor assessments from CT or MRI scans will be used to determine an objective response rate.
Progression-free survival | Baseline to 3 years
  Time to progressive disease
Number of patients with progression-free survival at 6 months | 6 months after the last cycle of treatment completed
  The percentage of patients with progression-free survival in the study
Overall survival | Baseline to 3 years
  Length of patient survival after starting study treatment
Measurement of TRC105 concentrations | Collected approximately every 63 days (3 cycles)
  Serum TRC105 concentrations will be measured using validated enzyme-linked immunoassay testing that will assist in analyzing the pharmacokinetics of the drug.
Measurement of TRC105 anti-product antibodies | Collected approximately every 63 days (3 cycles)
  Anti-product antibody concentrations will be measured using validated enzyme-linked immunoassay testing that will assist in analyzing immunogenicity.
Identify angiogenic protein biomarkers | Collected approximately every 63 days (3 cycles)
  A central reference lab will conduct biomarker testing that will assist in the analysis of the pharmacodynamics effects on circulating angiogenic biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Comprehensive Cancer Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided